CLINICAL TRIAL: NCT00246389
Title: Flexeril� (Cyclobenzaprine Hydrochloride) Community Based Study - An Evaluation of Cyclobenzaprine HCl Monotherapy and in Combination With Ibuprofen for Acute Back or Neck Muscle Pain With Muscle Spasm
Brief Title: An Effectiveness and Safety Study of Cyclobenzaprine HCl Alone or in Combination With Ibuprofen for Acute Back or Neck Muscle Pain With Muscle Spasm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002884
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Pain; Spasm
Keywords: muscle spasm; cyclobenzaprine hydrochloride
MeSH Terms: conditions — Pain; Spasm | interventions — cyclobenzaprine

INTERVENTIONS:
Drug: cyclobenzaprine hydrochloride

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of cyclobenzaprine HCl 5 mg (muscle spasm medication) taken three times a day, alone or in combination with ibuprofen 400 mg or 800 mg (pain relief medication) taken three times a day, for the treatment of back or neck muscle pain with muscle spasm.

DETAILED DESCRIPTION:
The objective of this multicenter, randomized, open-label, parallel-group, one-week study is to evaluate the effectiveness and safety of cyclobenzaprine HCl 5 mg three times a day for one week, alone or in combination with ibuprofen 400 mg or 800 mg taken three times a day, for acute back or neck muscle pain with muscle spasm. The primary measurement of efficacy is the subject-rated global impression of change after seven days of treatment, compared to baseline. Safety assessments during the study include the monitoring of adverse events, and a physical examination, assessment of vital signs and medical history of any present illnesses conducted during the baseline visit. The study hypothesis is that there will not be a statistically significant difference in patient ratings of global impression of change, muscle spasm, muscle pain, medication helpfulness, and functional ability, between the cyclobenzaprine HCl monotherapy group versus the cyclobenzaprine HCl/ibuprofen 400 mg and cyclobenzaprine HCl/ibuprofen 800 mg groups, for the treatment for acute back or neck muscle pain with spasm. Patients receive cyclobenzaprine HCl 5 mg administered orally three times a day for one week, or cyclobenzaprine HCl 5 mg with ibuprofen 400 mg administered orally three times a day for one week, or cyclobenzaprine HCl 5 mg with ibuprofen 800 mg administered orally three times a day for one week.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing neck or back pain for no more than 14 days
* Physician rating of the muscle spasm of the neck or back region as mild, moderate or severe
* Ability to discontinue all muscle relaxants, NSAIDs (anti-inflammatory drugs) and pain relievers, other than the study medications during the 7-day treatment period. (Cardioprotective doses of aspirin (<= 325 mg / day) may be taken.)

Exclusion Criteria:

* History of physician-diagnosed musculoskeletal neck or back muscle spasms within 12 months prior to the study
* neck or back pain radiating into the arms or legs
* history of serious medical conditions
* taken a narcotic or muscle relaxant within 12 hours of the baseline physician visit
* allergies to aspirin, NSAIDs or cyclobenzaprine HCl.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Subject-rated global impression of change from baseline, after seven days of treatment

SECONDARY OUTCOMES:
Subject global impression of change after 3 days; Proportion of responders after 3 and 7 days, Change from baseline in subject-rated pain intensity, muscle spasm intensity, functional ability, and medication helpfulness after 3 and 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Childers MK, Borenstein D, Brown RL, Gershon S, Hale ME, Petri M, Wan GJ, Laudadio C, Harrison DD. Low-dose cyclobenzaprine versus combination therapy with ibuprofen for acute neck or back pain with muscle spasm: a randomized trial. Curr Med Res Opin. 2005 Sep;21(9):1485-93. doi: 10.1185/030079905X61938. PMID 16197668